CLINICAL TRIAL: NCT04754165
Title: Postoperative Virtual Reality (VR) for Recovery After Bariatric Surgery
Brief Title: Postoperative VR for Recovery After Bariatric Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Israel-United States Binational Industrial Research and Development Foundation (Unknown); XRHealth (Unknown)
Responsible Party: Principal Investigator, Brian O'Gara, Assistant Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P001149
Record Dates: First submitted 2021-01-29; First posted 2021-02-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Bariatric Surgery Candidate; Postoperative Pain; Postoperative Complications
Keywords: Virtual Reality; ERAS
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Research participants will be randomized to one of two groups: immersive VR plus ERAS, or ERAS alone in a 1:1 allocation.
  The first 6 patients enrolled will be assigned to the VR group for the purposes of a pilot phase with the objective of identifying and refining any issues with the intervention. Data for these patients will not be included in the statistical analysis.
Who Masked: Outcomes Assessor
Masking Description: Assessors of the QOR15 recovery scale will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immersive Virtual Reality plus the enhanced recovery after surgery protocol (Experimental): Patients in the immersive VR group will don a VR headset connected to a software platform on a tablet, as well as noise cancelling headphones in the post anesthesia care unit (PACU) after surgery. Patients can choose their desired experience within the VR software from a selection of immersive environments and/or video content. Examples include sitting in a canoe on a river, on a peaceful meadow or in a forest. Patients also have the option to listen to guided meditation or select from a library of videos to watch on a web-based user interface.
  Patients in the VR group will also be treated according to the existing enhanced recovery after surgery protocol.
  Interventions: Other: Virtual Reality Immersive Relaxation
- Enhanced recovery after surgery protocol (No Intervention): Subjects in the control group will only undergo standard enhanced recovery after surgery care.

INTERVENTIONS:
Other: Virtual Reality Immersive Relaxation — The VR software developed allows patients to select from scenery such as mountains, the beach or from a selection of short videos, which are intended to promote relaxation.
  Arms: Immersive Virtual Reality plus the enhanced recovery after surgery protocol

SUMMARY:
The objective of this study is to investigate whether the addition of immersive virtual reality (VR) in the immediate postoperative period to an enhanced recovery after surgery (ERAS) protocol could improve postoperative recovery from bariatric surgery.

DETAILED DESCRIPTION:
The investigators propose conducting a randomized, controlled, single-center clinical trial of patients recovering from laparoscopic bariatric surgery. The objective is to investigate whether the use of virtual reality (VR) during the immediate postoperative period could improve patient reported quality of recovery and potentially reduce opioid analgesic requirements as compared to an existing ERAS protocol.

The investigators hypothesize that immersive VR will improve subjective quality of recovery scores at time of Post Anesthesia Care Unit (PACU) discharge as compared to standard ERAS.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing laparoscopic bariatric surgery at BIDMC under general anesthesia.

Exclusion Criteria:

* Age<18
* Open wounds or active infection of the face or eye area
* History of seizures or other symptom linked to an epileptic condition
* Patients with hearing aids who are unable to tolerate wearing headphones with their hearing aids
* Patients with a pacemaker or other implanted medical device
* Droplet or airborne precautions (as determined by BIDMC infection control policy)
* Non English Speaking or non Spanish Speaking
* Chronic opioid dependence (existing oral opioid prescription for >3 months, methadone, suboxone)

Drop Out Criteria: (after enrollment and randomization, before intervention)

- Surgery is converted to an open procedure (laparotomy), the patient will be withdrawn from the study as these patients are treated in a manner that is different than standard ERAS protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery Questionnaires (QoR-15) | Measured at time of post anesthesia care unit discharge, on average of 1 to 5 hours after surgery.
  The primary outcome of this study will be patient reported quality of recovery at time of PACU discharge, as assessed by the QOR-15. The QOR-15 is a validated instrument to assess postoperative recovery from the patient's perspective, assessing overall well-being, nausea, pain, and anxiety and depression following surgery.

SECONDARY OUTCOMES:
PACU Opioid Requirements | Measured throughout a patient's stay in the post anesthesia care unit, on average 1 to 5 hours after surgery.
  The postoperative opioid requirements following the patients surgery, will be measured in milligrams and converted to morphine dose equivalents.
Length of PACU stay | Duration of the patient's stay in the post anesthesia care unit, from time of admission to time of readiness for PACU discharge, on average 1 to 5 hours.
  The length of the patients stay in the Post Anesthesia Care Unit will be measured in minutes.
PACU pain scores using numeric rating scale | Administered every hour following admission to the post anesthesia care unit until discharge from the post anesthesia care unit, on average 1 to 5 hours.
  Clinically documented pain scores will be recorded on a scale from 0 (best outcome) to 10 (worst outcome).
Postoperative Quality of Recovery Questionnaires (QoR-15) score | Measured at 24 hours after post anesthesia unit discharge.
  The QOR-15 is a validated instrument to assess postoperative recovery from the patient's perspective, assessing overall well-being, nausea, pain, and anxiety and depression following surgery.
Hospital length of stay | Measured throughout the patients stay at the hospital, on average 1 to 3 days.
  The length of the patients stay following surgery.
Opioid requirements | Measured throughout the patients stay at the hospital, on average 1 to 3 days.
  Opioid requirements throughout the hospital stay.
Opioid-related adverse effects | Measured throughout the patients stay at the hospital, on average 1 to 3 days.
  Opioid-related adverse effects such as nausea or ileus.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P O'Gara, MD,MP, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espinosa-Leon JP, Mathura R, Chen G, Joseph M, Sadhwani T, Beydoun N, Hernandez ER, Riley T, Goodspeed V, O'Gara BP. Postoperative virtual reality for recovery after bariatric surgery: study protocol for a randomised clinical trial. BJA Open. 2024 Feb 5;9:100258. doi: 10.1016/j.bjao.2024.100258. eCollection 2024 Mar. PMID 38333728